CLINICAL TRIAL: NCT07141875
Title: Optimization Strategies for Pediatric Vaccination Scheduling in China: The Impact of Local Policies, Caregivers, Vaccination Staff, and the Cost-Effectiveness of Simultaneous and Combined Vaccinations
Brief Title: Child Vaccination Scheduling in China
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government); MSD China Holding Co Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB00001052-25094
Record Dates: First submitted 2025-08-15; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Vaccination Behavior
Keywords: Children vaccine; Simultaneous vaccination; Combination vaccines

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- • Caregiver of Children: Interviewees are parents or grandparents of children aged between 6 to 59 months.
  Interventions: Other: No intervention
- Vaccination and health care personnel: Interviewees are vaccination and health care personnel in each study site.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study without any interventions.

SUMMARY:
This study aims to optimize pediatric vaccine scheduling in China . The first objective is to gather information on current vaccine schedules in China. The second objective is to evaluate the impact of simultaneous vaccination and combination vaccines on costs and vaccination rates through feedback from caregivers and vaccination staff.

DETAILED DESCRIPTION:
The first objective will comprehensively collect vaccination programs for children under 6 years old in all 31 provinces of China (excluding Hong Kong, Macau, and Taiwan), covering both NIP and non-NIP vaccines that are suitable for children. The second objective is to evaluate the impact of simultaneous vaccination and combination vaccines on costs and vaccination rates. This will involve analyzing vaccination coverage for simultaneous vaccines across different regions in China, as well as assessing caregivers' perspectives on simultaneous vaccination, including their willingness, preferences, and factors influencing their vaccination decisions. Additionally, the study will explore vaccination staff attitudes, recommendation behaviors, and their reasons for recommending simultaneous and combination vaccines. For the survey, the sample will consist of caregivers of children (aged between 2 to 59 months) from 10 representative provinces/municipalities/autonomous regions as well as vaccination staff from institutions in the respective regions.

ELIGIBILITY:
Inclusion Criteria:

- For caregivers of children

* Children aged ≥2 months and ≤59 months
* Caregivers informed consent obtained For vaccination staff
* All vaccination staff currently working at the selected community health service centers or township health clinics on the day of the survey For retrospective analysis
* Children aged 5 years and under; with complete vaccination records. Complete vaccination records refer to a child having received all vaccines required by the NIP for their age group, with accurate dates recorded for each vaccination dose.

Exclusion Criteria:

- For caregivers of children

* Caregivers who are unable to participate in the survey due to physical or other objective reasons
* Caregivers with communication barriers
* Caregivers who do not consent to participate in the survey For vaccination staff
* Vaccination staff who do not consent to participate in the survey For retrospective analysis
* Children whose vaccination records are missing or incomplete
* Children whose vaccination has been delayed or not received due to medical contraindications.

Min Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample will consist of 6,000 caregivers of children (aged between 2 to 59 months) from 10 representative provinces/municipalities/autonomous regions as well as Vaccination and health care personnel in each study site.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
The economic value of optimized vaccination scheduling strategies | 2025.08-2025.09
  This study will comprehensively collect vaccination programs for children under 6 years old in all 31 provinces of China (excluding Hong Kong, Macau, and Taiwan), covering both NIP and non-NIP vaccines that are suitable for children.
  The economic value of optimized vaccination scheduling strategies with simultaneous vaccination and combination vaccines will be assessed using a cost-minimization and budget impact model with inputs collected in this study. The optimized vaccination scheduling strategie will be collected in this study through a literature review, a cross-sectional caregiver survey, a survey among vaccination staff, and an observational time and motion chart among the latter population.
Caregivers' willingness to simultaneous vaccination and combined vaccines | 2025.08-2025.09
  To evaluate the acceptance and willingness of different vaccination strategies, the survey will collect caregivers' knowledge, attitudes, and preferences on optimized vaccine scheduling strategies including simultaneous vaccination and combination vaccines, as well as factors influencing their decisions , such as the vaccination status of siblings of other children and elderly family members over 60 years old. The primary outcome variable will be willingness to simultaneous vaccination and combined vaccines, assessed using a 5-point ordinal scale (from "very unwilling" to "very willing").
Immunization records and vaccination coverage | 2025.08-2025.09
  Using data collected from children's immunization records, a retrospective analysis will explore how previous simultaneous vaccination behaviors affect their vaccination rate. By comparing the vaccination rates at different ages between children receiving vaccines concomitantly vs. separately and children who uses combination vaccines vs. single vaccines, the study will evaluate whether the optimized vaccine scheduling strategies including simultaneous vaccination and combination vaccines have an impact on children's vaccination coverage.

SECONDARY OUTCOMES:
Recommendation to simultaneous vaccination and combined vaccines | 2025.08-2025.09
  A survey will be used to evaluate the attitudes and recommendation behaviors among vaccination staff towards optimized vaccine scheduling strategies including simultaneous vaccination and combination vaccines. The outcome variable will be recommendation behavior, assessed on a 5-point Likert scale ranging from "strongly recommend" to "strongly not recommend". To examine the perceived difficulty of vaccine scheduling, the survey will collect potential contributing factors: complexity of immunization schedules, inaccuracy of manual scheduling, limited implementation of simultaneous vaccination strategies, insufficient use of combination vaccines, high demand for catch-up vaccination, and lack of clear guidance for non-NIP vaccines.
Vaccine hesitancy | 2025.08-2025.09
  Questions were designed in the questionnaire to evaluate the degree of vaccine hesitancy of interviewees. Respondents will be asked abound their confidence, convenience and complacency about vaccination of different non-NIP vaccines, so as to further explore the influencing factors of people's vaccination behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Health Science Center, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No